CLINICAL TRIAL: NCT05940740
Title: Investigation of the Effect of Training on the Side Effects of Chemotherapy Given Via the Mobile Health Application on the Quality of Life in Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NESLISAH YASAR KARTAL (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor-Investigator, NESLISAH YASAR KARTAL, Lecturer, University of Beykent
Organization: University of Beykent (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022.10.13-34
Record Dates: First submitted 2023-04-14; First posted 2023-07-11 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Mobile Phone Use; Nurse's Role
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Cell Phone Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERFERENCE (EXPERIMENT) (Experimental): 1. Giving patients with colorectal cancer about 20-30 minutes of training during chemotherapy with the mobile health application and answering face-to-face questions about the use of mobile health application.
  2. Sending a reminder message about the use of mobile health application via phone once a week. Answering the questions about the mobile health application and the training given during the chemotherapy application every two weeks / summarizing the training
  Interventions: Other: Colorectal-Mobile application
- CONTROL (No Intervention): 1. Giving approximately 20-30 minutes of routine treatment and care and answering questions during premedication application to colorectal cancer patients when they come to the unit to receive 1st cure chemotherapy.
  2. Pre-test-post-test at the beginning of the 1st course of treatment and at the end of the 3rd cycle of treatment

INTERVENTIONS:
Other: Colorectal-Mobile application — The use of Colorectal-Mobile application by the patients on a daily basis by the researcher will be monitored remotely via the management platform of the usage status of the mobile health application.
  Arms: INTERFERENCE (EXPERIMENT)

SUMMARY:
The incidence of colorectal cancer ranks fourth worldwide after lung, prostate and breast cancers. Although chemotherapy has an important place in the treatment of colorectal cancers, it can cause side effects such as diarrhea and fatigue in patients. Cancer patients' ability to cope with treatment side effects can be benefited from technological developments. Studies have shown that mobile health applications reduce symptom experience and increase quality of life in patients with breast cancer and leukemia.

DETAILED DESCRIPTION:
The incidence of colorectal cancer ranks fourth worldwide after lung, prostate and breast cancers. Although chemotherapy has an important place in the treatment of colorectal cancers, it can cause side effects such as diarrhea and fatigue in patients. Cancer patients' ability to cope with treatment side effects can be benefited from technological developments. Studies have shown that mobile health applications reduce symptom experience and increase quality of life in patients with breast cancer and leukemia. This research was planned as a quasi-experimental study with a pre-test-post-test control group in order to examine the effects of the mobile health application developed according to the Self-Care Disability Theory and the training given for chemotherapy side effects on the quality of life of colorectal cancer patients. The sample of the study will consist of patients who underwent chemotherapy outpatient (23 intervention group and 23 control group) with the diagnosis of colorectal cancer in the Internal Medicine Medical Oncology outpatient clinic of Istanbul University-Cerrahpasa Cerrahpasa Medical Faculty. Simple random sampling method, which is one of the probabilistic sampling methods, will be used to determine the intervention and control groups. Data will be obtained (pre-test) with the Patient Information Form, the Self-Care Needs Assessment Form, the Nightingale Symptom Assessment Scale (N-SDS), and the Cancer Treatment Functional Assessment-Colorectal Scale (FACT-C). Training will be provided to the initiative group through the mobile health application. Symptom management and quality of life will be evaluated by using data collection tools after the 1st and 2nd cycles of chemotherapy in intervention group patients. A face-to-face meeting with the initiative group is planned every two weeks. Once a week, an message will be sent to the intervention group patients reminding them to use the mobile health application. Control group patients will continue to receive routine treatment and follow-up. A post-test will be applied to the intervention and control groups in the third month (12 weeks after the first interview). In this study, it is aimed to compare the effectiveness of routine treatment and care with the use of a mobile health application developed according to the Self-Care Insufficiency Theory, considering the developments in today's technology, and to evaluate the effects of the two methods on the control of symptoms that may occur due to chemotherapy side effects in colorectal cancer patients and their care needs.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy was started with the diagnosis of colorectal cancer,
* Receiving adjuvant chemotherapy,
* His psychological and general condition is suitable for the interview and
* Identified as colorectal cancer patients who volunteered to participate in the study

Exclusion Criteria:

* Not diagnosed with colorectal cancer
* Not diagnosed adjuvant chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Colorectal | Two weeks
  The Functional Assessment of Cancer Therapy-Colorectal Scale was first developed by Ward et al. in 1999 in the USA by the Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System.
  The scale consists of a total of 5 dimensions and a total of 46 items. The scale consists of Ordinary Physical Status sub-dimension, Social Life and Family Status sub-dimension, intense Status sub-dimension, Activity Status sub-dimension and Other Concerns sub-dimensions.
  In the evaluation made with the FACT-C Scale, the subject is asked to answer each statement by observing the last 7th day indicator. Each item of the scale is evaluated on a 5-point Likert-type scale ("never" = 0, "very little" = 1, "some" = 2, "quite" = 3, "a lot" = 4). Its total score is between 0-136.
Patient Information Form | Two weeks
  The Patient Information Form was prepared considering the factors that may affect the self-care of patients diagnosed with colorectal cancer who underwent outpatient chemotherapy within a year. This form consists of a total of 19 questions questioning the characteristics of the individual, the disease and the treatment.
Nightingale Symptom Evaluation Scale | Two weeks
  The Nightingale Symptom Evaluation Scale (2009) was developed by Can and Aydıner for patients diagnosed with cancer. The scale includes three sub-dimensions. These sub-dimensions are "Physical Well-Being", "Social Well-Being" and "Psychological Well-Being".
  The answers given by the patients to the scale are scored from 0 to 4 and answered on a five-point Likert type scale. Patients are asked to evaluate these questions by choosing one of the points "No" "0 points", "Very little" "1 point", "A little" "2 points", "Quite" "3 points", "Too much" "4 points".

SECONDARY OUTCOMES:
Self-Care Needs Evaluation Form | Two weeks
  There are 28 statements in the Self-Care Needs Evaluation Form, which include the self-care needs of patients with colorectal cancer. In this form, it will question the self-care needs of colorectal cancer patients in case of universal, developmental and health deviations. Patients are asked to answer these statements by choosing one of the options "Yes", "Sometimes" or "No".

CONTACTS AND LOCATIONS:
Locations (1):
- Beykent University, Istanbul, Buyukcekmece, Turkey (Türkiye)